CLINICAL TRIAL: NCT01382628
Title: Determination of the Pathophysicologic Collagen Changes in the Diabetic Achilles Tendon.
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Paul J. Kim, DPM, Associate Professor, Dept of Plastic Surgery Director of Research, Georgetown University
Other Study IDs: 2011-101
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Diabetic Foot Ulcers; Equinus Deformity
Keywords: Diabetes; Ulcers; Equinus Deformity; Amputation; Achilles Tendon; Limb Loss
MeSH Terms: conditions — Diabetic Foot; Equinus Deformity; Diabetes Mellitus; Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A tissue sample (20mg) of the Achilles tendon will be collected at this time. This tissue will be preserved in a dry ice container and shipped to Midwestern University for processing by the sub-investigator (CC). The specimens will be labeled numerically with a predetermined subject number. No patient identifying information will be on these samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Preulcerative plantar foot lesion: An area on the plantar foot, usually at the location of a bony prominence, that presents with erythema, significant hyperkeratosis, or thin, shiny skin.
- Plantar ulcer no history of amputation: Plantar ulceration without a history of amputation or require an amputation.
- Plantar ulcer and digital amputation: Plantar ulceration who will be undergoing a digital amputation.
- Plantar ulcer and transmet amputation: Plantar ulceration who will be undergoing a transmetatarsal amputation.
- Plantar ulceration and choparts: Plantar ulceration who will be undergoing Chopart's or more proximal amputation.

SUMMARY:
This is a pilot study examining tendon collagen, collagen cross-linking, and markers of tendon extracellular matrix metabolism in the Achilles tendon of diabetic patients with ulcerations and amputations of the lower extremity.

DETAILED DESCRIPTION:
Diabetes is a pandemic problem with catastrophic effects on the physical, psychological, and economic lives of patients and their families, and also places a significant burden on the healthcare system. Changes in the integumentary system lead to plantar foot ulcerations, which increase the risk of limb amputations and death. Specifically, limitation of ankle joint dorsiflexion (equinus deformity) has been implicated as a major deforming force in the development and chronicity of plantar foot ulcerations in the diabetic population. A better mechanistic understanding of the intrinsic changes in the diabetic Achilles tendon would assist in explaining and potentially preventing the development of chronic foot ulcerations due to an equinus deformity.

This study will evaluate the relationship between limb loss progression and changes seen in collagen metabolic markers in the diabetic Achilles tendon. This will be assessed by collecting Achilles tendon samples in subjects who are at various stages of ulcer development or limb loss and who also demonstrate an equinus deformity. All Achilles tendon samples will be collected at the time of the Achilles lengthening procedure. There will be five subject groups consisting of subjects who have been identified with: 1)preulcerative plantar foot lesion 2)plantar ulceration without a history of amputation or require an amputation 3) plantar ulceration who will be undergoing a digital amputation 4) plantar ulceration who will be undergoing a transmetatarsal amputation or 5) plantar ulceration who will be undergoing Chopart's or more proximal amputation. Further, systemic changes (vasculopathy, peripheral neuropathy, nephropathy) will also be correlated with the above. The independent variables are the following: 1) collagen metabolic markers and 2)systemic changes. The dependent variable is limb loss progression assessed categorically (5 groups).

The 5 phases of this study include:

* Phase 1- Eligibility Assessment. Type I and Type II diabetic patients who present to the Georgetown University Hospital Limb Salvage Center will be evaluated for inclusion into our study based on inclusion/exclusion criteria.
* Phase 2- Interview and examination. Subjects will complete a comprehensive medical history, physical exam, and blood work (per Standard of Care. The PI or SI will perform an ankle joint range of motion examination and a Semmes-Weinstein 5.07 monofilament examination (per Standard of Care. A comprehensive metabolic panel will be ordered including hemoglobin A1C, BUN, and CR (per Standard of Care). Patients will then be referred to the vascular surgery department for noninvasive and/or invasive vascular studies (per standard of care) and patient will be scheduled for surgery at this time.
* Phase 3- Surgery and Tissue Collection. Surgery will be performed that may include ulcer debridement, soft tissue or bone reconstruction, or amputation (per SOC- only patients who have been identified as demonstrating an equinus deformity and agree to an Achilles tendon lengthening procedure along with ulcer debridement, or soft tissue or bone reconstruction, or amputation will be included in this study. Achilles tendon lengthening is considered an adjunctive SOC procedure in the surgical management of the diabetic foot). All subjects will have an Achilles tendon lengthening procedure performed by the primary (PK) or sub-investigators (JS and CA). A tissue sample (20mg) of the Achilles tendon will be collected at this time. This tissue will be preserved in a dry ice container and shipped to Midwestern University for processing by the sub-investigator (CC). The specimens will be labeled numerically with a predetermined subject number. No patient identifying information will be on these samples.
* Phase 4- Tissue and Data Processing. Assays will be performed on the tissue samples to measure specific metabolic markers of the diabetic Achilles tendon. Tendon collagen concentrations will be determined via quantification of the collagen specific amino acid, hydroxyproline by high performance liquid chromatography (HPLC) and fluorometric detection. The extent of collagen cross-linking will be determined by measuring the amount of pyridinium cross-link hydroxylysylpyridinoline will also be assessed though HPLC. RT-PCR will also be performed to determine the expression of various MMPs and TIMPs. The blood markers will be processed at Georgetown University Hospital. The Department of Vascular Surgery at Georgetown University will perform the noninvasive and invasive studies and the results of their findings will be reported to the investigators.
* Phase 5-Data Analysis. The results from the physical examination, laboratory studies, vascular studies, and tissue assays will be collected and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Type I or Type II Diabetes - diagnosed by their primary care provider
* Demonstrates an equinus ankle deformity - Less than 0 degrees of passive dorsiflexion at the ankle joint with the knee extended or flexed.
* Preulcerative plantar foot lesions - In the form of a callus with the epithelium intact

OR may also have the following:

* Plantar ulceration without a history of amputations
* Plantar ulceration with a history of digital amputations - or planned digital amputation
* Plantar ulceration with a history of transmetatarsal amputations - or planned transmetatarsal amputation
* Plantar ulceration with a history of Chopart's or more proximal amputation - or planned Chopart's or more proximal amputation

Exclusion Criteria:

* Does not demonstrate an equinus ankle deformity
* Cannot undergo elective surgery for any reason
* History of Achilles tendon lengthening procedure performed
* History of traumatic (acute or chronic) injury to the Achilles tendon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Georgetown University Hospital, Center for Wound Healing or patients admitted to the Georgetown University Hospital (where the Limb service has been designated as a consulting or primary service) will be recruited into the study. Patients scheduled for an Achilles tendon lengthening procedure (as part of their SOC) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Structural and metabolic changes | 1 year
  Characterize the structural and metabolic changes in the diabetic Achilles tendon as related to limb loss.

SECONDARY OUTCOMES:
Relationship between collagen changes and system changes | 1 year
  Describe the relationship between collagen changes and system changes in the diabetic patient.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Kim, DPM, Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital Center for Wound Healing, Washington D.C., District of Columbia, United States